CLINICAL TRIAL: NCT06694116
Title: Charcoal Carbon Black Dye Use in Sentinel Lymph Node Mapping in Early Stage Vulvar Cancer
Acronym: IFLND
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Mustafa Albayrak, Principal Investigator, Istanbul University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2024/1551
Record Dates: First submitted 2024-11-15; First posted 2024-11-19 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-11

CONDITIONS: Vulval Cancer; Sentinel Lymph Node Detection
Keywords: vulvar cancer; observatinal study; charcoal carbon dye
MeSH Terms: conditions — Vulvar Neoplasms

STUDY DESIGN:
Intervention Model Description: The aim of this single arm prospective observational and intervational study is to investigate the detection rate, sensitivity, specificity, negative predictive value and positive predictive value of using charcoal carbon dye as a sentinel tracer in IFLN basin. Early stage primary vulvar tumors less than 4 cm with any histology but without any clinically or radiographically detectable inguinofemoral lymph nodes will be included. The parameters will be compared to pathologic results obtained from full IFLND.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single arm study using carbon dye as a sentinel lymph node agent in early vulvar cancer (Experimental): Single arm study using carbon dye as a sentinel lymph node agent in early vulvar cancer. Sterile charcoal carbon dye will be injected around vulvar tumor which will be searched in IFLND. No other arms.
  Interventions: Diagnostic Test: sentinel lymph node biopsy using carbon dye

INTERVENTIONS:
Diagnostic Test: sentinel lymph node biopsy using carbon dye — Sterile Charcoal carbon dye peritumoral injection will be performed around vulvar tumor and inguinofemoral lymph node dissection will be done 20 min later (unilateral or bilateral)

SUMMARY:
The aim of this study is to investigate the detection rate, sensitivity and specifity of charcoal carbon black dye as a sentinel lymph node tracer in inguinofemoral lymph node(s) in early stage vulvar cancer

DETAILED DESCRIPTION:
Vulvar cancer is a rare malignancy constituting approximately only 4% of all gynaecological malignancies. Treatment depends on histopathology and stage with surgery being the primary treatment modality in early stages with or without adjuvant radiotherapy depending on tumor margin status and involvement of inguinofemoral lymph nodes. Bilateral or unilateral surgical evaluation of inguinofemoral lymph nodal basin is an important part of the surgical procedure in early stage disease besides vulvar surgery since metastatic involvement dramatically changes stage, adjuvant treatment and surveillance. The usual method for surgical evaluation of inguinofemoral lymph nodes is full inguinofemoral lymph node dissection (IFLND). However, IFLND is highly related to complications such as lymphedema, incisional detachment, lymphocyst formation, lymphangitis, vessel injury and deep venous thrombosis. Over the last 10-15 years sentinel lymph node biopsy of inguinofemoral lymph nodes became a well-accepted form of surgical evaluation procedure instead of IFLND.

The present guidelines offer sentinel lymph node biopsy using various tracers and dyes used alone or in combination (either a blue dye or indocyanine green -ICG (indocyanine green) - is offered in addition to radiocolloid tracer). However, radiocolloid and ICG tracers requires expensive equipment and cumbersome procedures. On the contrary, sterile charcoal carbon dye is inexpensive and does not necessitate any further equipment to be detected. It is actually used to mark the point of resection of colon during colorectal surgery by general surgeons which is injected to the colonic mucosa preoperatively by colonoscopy.

The aim of the present study is to investigate the sensitivity, specificity, negative predictive value and positive predictive value of using charcoal carbon dye as a sentinel tracer in IFLN basin. Early-stage primary vulvar tumors less than 4 cm with any histology but without any clinically or radiographically detectable inguinofemoral lymph nodes will be included into study. Peritumoral four quadrant injections of carbon dye each 0.5 cc or two injections of 3 and 9 o'clock each 1 cc will be given. Following a 20 min interval inguinofemoral area will be dissected and full lymphadenectomy will be performed irrespective of sentinel lymph node recovery since bilateral or unilateral full inguinofemoral lymph node dissection is done in the department of the study so far. Detection rate and other parameters (sensitivity, specificity and etc.) will be compared to results of pathologic evaluation of full IFLND.

Investigators are currently two ongoing studies using charcoal carbon dye as a sentinel tracer to investigate its effectiveness compared to ICG (one in endometrial cancer and the other in ovarian cancer). Both studies are registered to ClinicalTrials.gov (NCT06163963 and NCT05927818). This will be the third of the study series using charcoal carbon dye as sentinel lymph node mapping method in gynecologic cancers (Forth one will be registered in ClinicalTrials.gov shortly in cervical cancers compared to ICG).

ELIGIBILITY:
Inclusion Criteria: Women with primary early stage vulvar cancer (Figo stage I and II) who will be operated with vulvar and inguinofemoral dissection -

Exclusion Criteria: Women less than 18 years of age or who declines surgery

-

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — women with vulvar cancer
Enrollment: 40 (Estimated)
Dates: Start 2024-05-30 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Detection rate of sentinel lymph node(s) | Two years
  Detection of sentinel lymph node for both unilateral or bilateral inguinofemoral region (in percentages). (For instance: In what percentage a unilateral or bilateral sentinel lymph node stained with carbon dye - either negative or positive - is detected?)
Sensitivity of sentinel lymph node mapping | Two years
  Sentinel lymph nodes true positive for malignancy in percentages divided by all sentinel lymph nodes either positive or negative for malignancy which is determined by pathologic report after all full inguinofemoral lymph nodes are examined for malignancy
Specifity of sentinel lymph node mapping | Two years
  Detection of true negative sentinel lymph nodes for malignancy divided by all sentinel lymph nodes either positive or negative for malignancy which is determined after all full inguinofemoral lymph nodes are examined pathologically
Negative and positive predictive values | Two years
  Detection of ratio of negative and positive for malignancy with sentinel lymph nodes to negative and positive for malignancy detected by full inguinofemoral lymph node dissection respectively

CONTACTS AND LOCATIONS:
Overall Officials: Yavuz Salihoglu, Prof. Dr., Study Director — ISTANBUL UNİVERSİTY MED FAC DEPT. OF OBSTET AND GYNECOL. DIVISION OF GYNECOLOGİC ONCOLOGY
Locations (1):
- Istanbul University Med Fac Dept. of Obstet and Gynecol. Division of Gynecologic Oncology, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be available in two years and will be in available forever.
Access Criteria: All data set and results will be planned to open, no criteria.

REFERENCES:
- [Background] Holloway RW, Abu-Rustum NR, Backes FJ, Boggess JF, Gotlieb WH, Jeffrey Lowery W, Rossi EC, Tanner EJ, Wolsky RJ. Sentinel lymph node mapping and staging in endometrial cancer: A Society of Gynecologic Oncology literature review with consensus recommendations. Gynecol Oncol. 2017 Aug;146(2):405-415. doi: 10.1016/j.ygyno.2017.05.027. Epub 2017 May 28. PMID 28566221
- [Background] ASGE Technology Committee; Kethu SR, Banerjee S, Desilets D, Diehl DL, Farraye FA, Kaul V, Kwon RS, Mamula P, Pedrosa MC, Rodriguez SA, Wong Kee Song LM, Tierney WM. Endoscopic tattooing. Gastrointest Endosc. 2010 Oct;72(4):681-5. doi: 10.1016/j.gie.2010.06.020. PMID 20883844
- [Background] Rychlik A, Bidzinski M, Rzepka J, Piatek S. Sentinel lymph node in vulvar cancer. Chin Clin Oncol. 2021 Apr;10(2):19. doi: 10.21037/cco-20-202. Epub 2020 Dec 11. PMID 33353362
- [Background] Penn CA, Schneiter MK, Watson CH. Sentinel Lymph Node Evaluation in Early-Stage Vulvar Cancer. Curr Treat Options Oncol. 2024 Jan;25(1):20-26. doi: 10.1007/s11864-023-01165-1. Epub 2024 Jan 3. PMID 38170388
- [Background] Pedrao PG, Guimaraes YM, Godoy LR, Possati-Resende JC, Bovo AC, Andrade CEMC, Longatto-Filho A, Dos Reis R. Management of Early-Stage Vulvar Cancer. Cancers (Basel). 2022 Aug 29;14(17):4184. doi: 10.3390/cancers14174184. PMID 36077719